CLINICAL TRIAL: NCT06279793
Title: Intravenous Fish Oil Based Lipid Emulsion to Enhance Recovery in High-Risk Cardiac Surgery Patients: a Phase II Multicenter Trial - A Randomized, Placebo-controlled Trial -
Brief Title: Intravenous Fish Oil Based Lipid Emulsion to Enhance Recovery in High-Risk Cardiac Surgery Patients
Acronym: MODIFY CSX
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GCP-Service International West GmbH (Industry)
Collaborators: University Hospital, Bonn (Other); University Hospital Muenster (Other); University Hospital Goettingen (Other); University Hospital Schleswig-Holstein (Other); Charite University, Berlin, Germany (Other); Wuerzburg University Hospital (Other); Johannes Gutenberg University Mainz (Other); University Hospital Augsburg (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MODIFY CSX
Record Dates: First submitted 2023-09-13; First posted 2024-02-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Intensive Care Unit; Coronary Artery Bypass Grafting (CABG); High Risk Patients; Cardiopulmonary Bypass; Elective Cardiac Surgery; Valvular Heart Surgery; Multiple Valve Surgeries; Combined Cardiac Procedures; Aortic Surgical Procedures
Keywords: intensive care unit; elective cardiac surgery; fish oil; medical nutrition therapy; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Fish Oils; fish oil triglycerides; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomization will be stratified by site, employing a web-based system using a 1:1 ratio to either intravenous fish oil-based lipid emulsion (Omegaven®), or placebo.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients as well as clinical staff and outcome assessors not involved in the study will be blinded to study intervention allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients will receive 0.20 g fish oil/kg BW/d (≙2 mL Omegaven®/kg BW/d).
  Interventions: Drug: Fish Oil
- Control group (Placebo Comparator): Patients will receive 0,9% NaCl in volume 2 mL/kg BW/d (placebo).
  Interventions: Drug: Intravenous 0.9% Sodium Chloride

INTERVENTIONS:
Drug: Fish Oil — Omegaven® is a 10% fish oil emulsion with a high percentage of long-chain n-3 fatty acids - mainly eicosapentaenoic acid and docosahexaenoic acid. It optimises the fatty acid pattern in parenteral nutrition and is a source of polyunsaturated n-3 fatty acids as cell membrane components and precursors for eicosanoids.
  Omegaven® is manufactured by Fresenius-Kabi, Germany and is available in 100 mL bottles for study purpose.
  Each 100 mL of Omegaven® contains 10 g of fish oil (0.1 g/mL).
  Timeframe: Day -1: 0.20 g fish oil/kg BW/d (the treatment should be started 24 to 3 h before surgery, can be given as 3-6 hours infusion); intraoperative day 0: no dose; postoperative day 0: 0.20 g fish oil/kg BW/d; postoperative days 1 to max. 7): 0.20 g fish oil/kg BW/d
  Other Names: Omegaven®
  Arms: Treatment group
Drug: Intravenous 0.9% Sodium Chloride — Intravenous 0.9% Sodium Chloride (volume 2 mL/kg BW/d) provided at the same timepoints as the intervention.
  Other Names: Saline Infusion
  Arms: Control group

SUMMARY:
The MODIFY CSX study is a prospective, randomized, placebo-controlled trial conducted in heart centers in Germany.

A total of 120 high-risk cardiac surgery patients will receive either 0.20 g fish oil/kg body weight (BW) + standard of care versus same volume of placebo (NaCl) + standard of care.

DETAILED DESCRIPTION:
The proposed hypothesis is that the therapeutic strategy tested in this randomized trial will decrease the occurrence of postoperative atrial fibrillation, which ultimately leads to faster time to discharge alive. This in turn significantly improves the patients' mid and long-term outcomes and dramatically reduces associated healthcare related costs.

Duration of intervention: until discharge from ICU, death or postoperative day 7 on ICU, whichever comes first.

Treatment Group: Patients will receive 0.20 g fish oil/kg BW/d (≙ 2 mL Omegaven®/kg BW/d).

Control Group: Patients will receive 0,9% NaCl in dose 2 mL/kg BW/d (placebo).

Follow-up per patient: at day 30, months 3, 6, and 12.

Primary endpoint (Phase II study):

The primary endpoint for this phase II clinical trial is be the onset and occurence of atrial fibrillation after cardiac surgery (AFACS) until day 7 after surgery (on ICU and normal ward).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to study participation
2. Adult patients (≥ 18 years)
3. Patients scheduled to undergo elective cardiac surgery with the use of CPB, who are defined as high risk based on having (i) one of the following surgical procedures: valvular heart surgery only, CABG, combined valve and CABG, multiple valve surgeries, combined cardiac procedures, aortic surgical procedures (aortic arch and/or descending aorta; aortic valve+ascending aorta) and (ii) at least one of the following additional risk factors: (a) a high perioperative risk profile, defined as predicted operative mortality of ≥8% (EuroSCORE II), (b) age ≥70, (c) Clinical Frailty Score 4 or more, (d) urgent surgery (defined as to be performed within 24-48 hours after admission), (e) left ventricular ejection fraction <35%

Exclusion Criteria:

1. Known hypersensitivity to fish oil/fish products or egg protein
2. Pregnancy or lactation period
3. Previous history of chronic atrial fibrillation, atrial flutter and/or atrial tachyarrhythmia
4. Inability or unwillingness of individual to give written informed consent
5. Not expected to survive an additional 48 hours from screening evaluation
6. Lack of commitment to full, aggressive care (anticipated withholding or withdrawing treatments in the first week but isolated "Do not Resuscitate" [DNR] acceptable)
7. Patients admitted with diabetic ketoacidosis or non-ketotic hyperosmolar coma
8. Patients receiving extracorporeal mechanical assist device (e.g. ECLS, or IABP) or advanced heart failure therapies (e.g. TAH, VAD)
9. Enrolment in anyinterventional trial within the last 30 days
10. Already receiving FO-containing medical nutrition products
11. Severe malnutrition (as defined by the BMI <18.5)
12. Severe liver dysfunction defined by Child Pugh Class C.
13. Severe chronic kidney dysfunction defined by the National Kidney Foundation (NKF) stage 4 and 5 by using the glomerular filtration rate (GFR <30ml/min)
14. Known severe coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation | Postoperative days 0-7
  The primary objective is to demonstrate superiority of fish oil compared to placebo in the prevention of atrial fibrillation until 7 days after surgery. This clinical endpoint is assessed as part of the clinical practice.

SECONDARY OUTCOMES:
Mechanical ventilation | Postoperative days 0-7, ICU discharge (approximately 3-4 days after surgery), hospital discharge (approximately 1-2 weeks after surgery), day 30 follow-up
  Duration of mechanical ventilation
Adverse Events | Preoperative day -1 to 12 months follow-up
  AEs leading to discontinuation/AEs at least possibly related to the IMP/SAEs
Delta Sequential Organ Failure Assessment Score (SOFA) Score | Postoperative days 0-7
  A scoring system that assesses the performance of several organ systems in the body (neurologic, blood, liver, kidney, and blood pressure/hemodynamics) and assigns a score based on the data obtained in each category.
Stroke | Postoperative days 0-7
  Incidence of stroke
Inotropics/vasopressors | Postoperative days 0-7, ICU discharge (approximately 3-4 days after surgery), hospital discharge (approximately 1-2 weeks after surgery), day 30 follow-up
  Duration of inotropic/vasopressor support
Acute Kidney Injury | Postoperative days 0-7
  Kidney Disease: Improving Global Outcomes [KDIGO] stages 1-3
Infection rate | Postoperative days 0-7
  Number of infections
Survival status | ICU discharge (approximately 3-4 days after surgery), hospital discharge (approximately 1-2 weeks after surgery), day 30 follow-up, months 3, 6, and 12 follow-up
  Overall survival
Quality of Life (SF-36) | Screening (preoperative day -7 until day -1), day 30 follow-up, 3, 6, and 12 months follow-up
  To measure the quality of life
Postoperative bleeding | Postoperative days 0-7
  Bleeding after surgery
ICU length of stay | ICU discharge (approximately 3-4 days after surgery)
  Number of days alive in the ICU
Hospital length of stay | Hospital discharge (approximately 1-2 weeks after surgery)
  Number of days alive in the hospital
Physical activity assessment | Screening (preoperative day -7 until day -1), day 30 follow-up, 3 and 6 months follow-up
  Katz activities of daily living (ADL) and Lawton's Instrumental ADL (IADL)
Days alive and out of hospital | Day 30 follow-up, 3, 6, and 12 months follow-up
  Time to be alive and discharge from hospital
Time to discharge alive | ICU discharge (approximately 3-4 days after surgery), hospital discharge (approximately 1-2 weeks after surgery)
  Time to be alive and discharged from ICU/hospital
Weaning from cardiopulmonary bypass (CPB) | Intraoperative day 0 (during surgery)
  Number of attempts to wean from CPB during surgery
Persistent Organ Dysfunction + Death | Postoperative days 0-7, ICU discharge (approximately 3-4 days after surgery), hospital discharge (approximately 1-2 weeks after surgery), day 30 follow-up
  Requiring supportive technologies during the convalescent phase of critical illness
ICU Readmission rates | Day 30 follow-up, 3, 6, and 12 months follow-up
  Readmission to ICU
Hospital Readmission rates | Day 30 follow-up, 3, 6, and 12 months follow-up
  Readmission to hospital

OTHER OUTCOMES:
Optional tertiary endpoint: Ultrasound measurement of thigh skeletal muscle mass | Screening (preoperative day -7 until day -1), ICU discharge (approximately 3-4 days after surgery), hospital discharge (approximately 1-2 weeks after surgery)
  Ultrasound measurement of thigh skeletal muscle mass
Optional tertiary endpoint: Functional Status Score for Intensive Care Unit (FSS-ICU) | Screening (preoperative day -7 until day -1), ICU discharge (approximately 3-4 days after surgery), hospital discharge (approximately 1-2 weeks after surgery)
  Functional Status Score for Intensive Care Unit (FSS-ICU)
Optional tertiary endpoint: Short Physical Performance Battery test (SPPB) | Screening (preoperative day -7 until day -1), ICU discharge (approximately 3-4 days after surgery), hospital discharge (approximately 1-2 weeks after surgery)
  Short Physical Performance Battery test (SPPB)
Optional tertiary endpoint: Hand grip/held dynamometer | Screening (preoperative day -7 until day -1), ICU discharge (approximately 3-4 days after surgery), hospital discharge (approximately 1-2 weeks after surgery)
  Hand grip/held dynamometer
Optional tertiary endpoint: Inflammatory response | Intraoperative day 0, postoperative days 0-7
  Inflammatory response and immune function as measured by markers of the clinical routine (e.g. IL6, IL10, CRP, white blood cell count [WBC], PCT, TNF-a)
Optional tertiary endpoint: Left ventricular ejection fraction | Preoperative day -1, hospital discharge (approximately 1-2 weeks after surgery), day 30 follow-up, 3 and 6 months follow-up
  Left ventricular ejection fractLeft ventricular ejection fractionion
Optional tertiary endpoint: Manual Muscle Testing (MMT) | Screening (preoperative day -7 until day -1), ICU discharge (approximately 3-4 days after surgery), hospital discharge (approximately 1-2 weeks after surgery)
  Manual Muscle Testing (MMT)
Optional tertiary endpoint: Vasoactive-Inotropic Score (VIS) | Postoperative days 0-7
  Vasoactive-Inotropic Score (VIS)
Optional tertiary endpoint: Therapeutic Intervention Scoring System (TISS) | Postoperative days 0-7
  A method for measuring workload and calculating costs in the ICU
Optional tertiary endpoint: Development of delirium | Postoperative days 0-7
  Assessed by the CAM ICU score
Optional tertiary endpoint: Hemodynamic parameters | Intraoperative day 0, postoperative days 0-7
  Adequate hemodynamic support, as defined by stable Cardiac Index, cardiac output (CO), Cardiac Power Index, mean arterial pressure (MAP), central vein pressure (CVP), pulmonary artery diastolic pressure (to be measured every 8 hours for first 72 hours post-op or until removal of pulmonary artery catheter, whatever comes first
Optional tertiary endpoint: Clinical frailty scale | Screening (preoperative day -1 until day -7), day 30 follow-up, 3 months follow-up
  A 9-point scale that quantifies frailty based on function in individual patients
Optional tertiary endpoint: Simplified Acute Physiology Score (SAPS) | Postoperative days 0-7
  Estimates the probability of mortality for ICU patients on admission
Optional tertiary endpoints: Further routine biomarkers | Intraoperative day 0, postoperative days 0-7
  Further routine biomarkers: creatinine, urea, bilirubin, troponin, triglycerides if available
Separate Sub-study | Preoperative day -1, intraoperative day 0, postoperative days 0-7, hospital discharge (approximately 1-2 weeks after surgery)
  Serial blood samples and - if available - tissue samples from patients (if these result from the routine surgical procedure) will be collected in concerning patients at the day before (only blood samples), during surgery (only tissue sample if available), and once daily after surgery while the patients are on ICU (only blood samples):
  * Specialized pro-resolving mediators (SPMs) and more specific markers of the inflammatory response, such as the production of leukotriene B5 (LTB5), leukotriene B4 (LTB4), 5-hydroxyeicosapentaenoic acid (5-HEPE) and production of 5-hydroxyeicosatetraenoic acid (5-HETE)
  * SPMs, such as maserins and resolvins
  * Oxidative stress (oxidative reduction potential, Malondialdehyde)
  * Membrane incorporation of PUFAs (white blood cells) &amp; tissue samples
  * Activation of survival kinases (such as extracellular-signal regulated

CONTACTS AND LOCATIONS:
Overall Officials: Christian Stoppe, Prof. Dr., Study Director — Wuerzburg University Hospital
Locations (8):
- Germany (8):
  - University Hospital Augsburg, Augsburg
  - Charité Universitätsmedizin Berlin, Berlin
  - University of Bonn, Bonn
  - University Hospital Goettingen, Göttingen
  - University Hospital Hamburg-Eppendorf, Hamburg
  - University Medical Center Schleswig-Holstein, Kiel
  - University Hospital Mainz, Mainz
  - University Hospital Muenster, Münster

IPD SHARING:
Plan to Share IPD: No